CLINICAL TRIAL: NCT06700265
Title: Ultrasound Airway Examination as a Tool for Detection of Difficult Intubation in Adult Patients
Status: Not yet recruiting | Type: Observational
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Other Study IDs: airway ultrasound
Record Dates: First submitted 2024-11-11; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Difficult Airway
Keywords: airway ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the goal of the observational study to measure the effectiveness of neck ultrasound in prediction of difficult intubation in adult patients

DETAILED DESCRIPTION:
All participant undergoing elective surgery under general anesthesia will go a detailed preoperative sonographic assessment by the anesthesiologist who has experience in airway ultrasound for measurement of Hyomental distance, thyrohyoid distance, thyroid cricoid, anterior soft tissue thickness at levels of hyoid bone, cricoid cartilage and vocal cord and all measurement will be measured in neutral and sniffing position.

after induction of general anesthesia intubation will done by macintosh laryngoscope and degree of difficulty of intubation will be measured by cormack-lehane classification without any external manipulation

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above18 years old
* Both sex
* Requiring general anesthesia with endotracheal intubation

Exclusion Criteria:

* Emergency surgery,
* patients with limited mouth, head or neck movement,
* patients with temporomandibular joint impairment,
* fracture or tumors of mandible,
* patients requiring awake intubation,
* uncooperative patients,
* any cervical spine limitation movement
* neck swelling or tumor
* Prominent teeth deformities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all population undergoining surgical operation requiring general anesthesia and endotracheal intubation
Sampling Method: Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
measurement of effectiveness of neck ultrasound use of ultrasound measurement in prediction of difficult intubation | 30 min after ultrasound measurements at time of induction of anesthesai
  In cormack lehan classification of laryngoscopy view

SECONDARY OUTCOMES:
Hyomental distance in neutral position | 30 min before operation
  In centimetres
Throhyoid distance in neutral position | 30 min before operation
  In centimetres
Cricothyriod distance in neutral position | 30 min before operation
  In centimetres
Anterior soft tissue thickness at level of hyoid bone in neutral position | 30 min before opeqrtio
  In centimetres
Anterior soft tissue thickness at level of epiglottis in neutral position | 30 min befor operation
  In centimetres
Anterior soft tissue thickness at level of vocal cord in neutral position | 30 min before operation
  In centimetres
Hyomental distance in sniffing position | 30 min before operation
  In centimetres
Thyrohyoid distance in sniffing position | 30 min before operation
  In centimetres
Cricothyroid distance in sniffing position | 30 minutes before operation
  In centimetres
Anterior soft tissue thickness at level of hyoid bone in sniffing position | 30 min before operation
  In centimetres
Anterior soft tissue thickness at level of epiglottis in sniffing position | 30 min before operation
  In centimetres
Anterior soft tissue thickness at level of vocal cord in sniffing position | 30 min before operation
  In centimetres

OTHER OUTCOMES:
Age | 30 min before operation
  Years

CONTACTS AND LOCATIONS:
Overall Officials: ayman ali ghoneim, MD in anesthesia, Study Director — national cancer institute in egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: for 1 year

REFERENCES:
- [Result] Parameswari A, Govind M, Vakamudi M. Correlation between preoperative ultrasonographic airway assessment and laryngoscopic view in adult patients: A prospective study. J Anaesthesiol Clin Pharmacol. 2017 Jul-Sep;33(3):353-358. doi: 10.4103/joacp.JOACP_166_17. PMID 29109635
- [Result] Roth D, Pace NL, Lee A, Hovhannisyan K, Warenits AM, Arrich J, Herkner H. Airway physical examination tests for detection of difficult airway management in apparently normal adult patients. Cochrane Database Syst Rev. 2018 May 15;5(5):CD008874. doi: 10.1002/14651858.CD008874.pub2. PMID 29761867
- [Result] Gomes SH, Simoes AM, Nunes AM, Pereira MV, Teoh WH, Costa PS, Kristensen MS, Teixeira PM, Pego JM. Useful Ultrasonographic Parameters to Predict Difficult Laryngoscopy and Difficult Tracheal Intubation-A Systematic Review and Meta-Analysis. Front Med (Lausanne). 2021 May 28;8:671658. doi: 10.3389/fmed.2021.671658. eCollection 2021. PMID 34124099